CLINICAL TRIAL: NCT04109092
Title: INtravesical Phase 1/1b Study of STING Agonist E7766 in NMIBC Including Subjects Unresponsive to BCG Therapy, INPUT-102
Brief Title: A Study of Stimulator of Interferon Genes (STING) Agonist E7766 in Non-muscle Invasive Bladder Cancer (NMIBC) Including Participants Unresponsive to Bacillus Calmette-Guerin (BCG) Therapy, INPUT-102
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: There was no enrolment of participants.Unscheduled Clinical Study Closure - Eisai Network Company Decision, November 12, 2020.
Sponsor: Eisai Inc. (Industry)
Collaborators: H3 Biomedicine Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: E7766-G000-102; 2019-000161-21 (EudraCT Number)
Record Dates: First submitted 2019-08-27; First posted 2019-09-30 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-07

CONDITIONS: Urinary Bladder Neoplasms
Keywords: E7766; Non-Muscle Invasive Bladder Cancer; Intravesical administration; Ta or T1 Papillary Disease; Stimulator of Interferon Genes Agonist; Carcinoma in situ; BCG Unresponsive
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms; Carcinoma in Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation: NMIBC And BCG Unresponsive NMIBC (Experimental)
  Interventions: Drug: E7766
- Dose Expansion: CIS With/Without Ta or T1 (Experimental)
  Interventions: Drug: E7766
- Dose Expansion: High-grade Ta or T1, Without CIS (Experimental)
  Interventions: Drug: E7766

INTERVENTIONS:
Drug: E7766 — E7766, solution, intravesically.

SUMMARY:
This is an open label, multicenter, phase 1/1b study to assess safety/tolerability and preliminary clinical activity of E7766 as a single agent administered intravesically in participants with NMIBC. Both intermediate risk and BCG-unresponsive NMIBC participants will be included.

DETAILED DESCRIPTION:
The Phase 1/1b study consist of two parts: Dose Escalation and Dose Expansion. In the Dose Escalation Part, E7766 will be administered intravesically to participants with intermediate risk NMIBC or participants with BCG unresponsive NMIBC with increased dose levels to assess safety/tolerability profile of E7766 and to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of E7766. In the Dose Expansion Part, E7766 at RP2D will be administered to participants with NMIBC with or without carcinoma in situ (CIS) to confirm safety and assess preliminary clinical activity of E7766 as a single agent. Clinical activity will be evaluated by complete response (CR) rates at 3 months, 6 months, 12 months, 18 months, 24 months, and by duration of complete response (DOCR) in all participants who have achieved CR on treatment with E7766.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
2. Life expectancy greater than (>) 2 years in the view of the investigator.
3. Participants must have biopsy proven transitional or predominantly transitional cell NMIBC.
4. For the Dose Escalation part of the study, the following participants will be included:

   1. Both, lower and higher dose escalation cohorts:

      Participants with intermediate risk NMIBC
   2. Only higher dose escalation cohorts:

   Participants with BCG Unresponsive NMIBC despite prior adequate treatment. Furthermore, all participants should be indicated for radical cystectomy as the standard of care for BCG unresponsive NMIBC. Participants who are undergoing radical cystectomy as well as participants who have refused to undergo radical cystectomy will be eligible to participate in the Dose Escalation part of the study. For participants who are undergoing radical cystectomy, date of surgery should not be delayed more than 3 months after Day 1 of dosing.

   For the Dose Expansion part of the study, the following participants will be included:

   Participants with histologically confirmed
   1. CIS (with or without concomitant non-muscle invasive, Ta or T1 papillary disease) (Arm 1) Or
   2. Non-muscle invasive high-grade Ta or T1 papillary disease without CIS (Arm 2) that is deemed to be unresponsive to BCG therapy despite prior adequate treatment. Furthermore, participants should be indicated for radical cystectomy as the standard of care for BCG unresponsive NMIBC but have refused to undergo radical cystectomy.

   Intermediate risk NMIBC: is defined as any participant with a high-grade Ta less than or equal to (<=) 3 cm or low-grade T1 tumor or with histologically confirmed multiple and/or recurrent low-grade Ta tumor with either 1 or 2 of the following 4 factors
   1. Multiple tumors
   2. Tumor >3 centimeter (cm)
   3. Early recurrence (less than [<] year)
   4. Frequent recurrences (>1 per year)

   BCG Unresponsive NMIBC is defined as being at least 1 of the following:
   1. Persistent or recurrent CIS alone or with recurrent Ta/T1 (noninvasive papillary disease/tumor invades the subepithelial connective tissue) disease within 12 months of completion of adequate BCG therapy.
   2. Recurrent high-grade Ta/T1 disease within 6 months of completion of adequate BCG therapy.
   3. T1 high-grade disease at the first evaluation following an induction BCG course

   Adequate BCG therapy is defined as at least 1 of the following:
   1. At least 5 of 6 doses of an initial induction course plus at least 2 of 3 doses of maintenance therapy.
   2. At least 5 of 6 doses of an initial induction course plus at least 2 of 6 doses of a second induction course.
5. Participants must consent to repeat biopsies to allow the acquisition of fresh formalin-fixed paraffin embedded (FFPE) material (obtained within 8 weeks prior to treatment initiation with E7766)
6. Participants must consent to repeat blood draws as indicated in the schedule of assessments.
7. Participant must consent to providing cystectomy tumor sample in the event that cystectomy is performed following treatment with E7766.
8. Immunosuppressive doses of systemic medications, such as steroids or absorbed topical steroids (doses >10 milligram per day (mg/d) prednisone or equivalent) must be safely discontinued at least 4 weeks before study drug administration.
9. Participants with prior Hepatitis B or C are eligible if they have adequate liver function.
10. Left ventricular ejection fraction (LVEF) >50 percent (%) on echocardiography or multiple gate acquisition (MUGA) scan.
11. Adequate renal function, bone marrow function and liver function.

Exclusion Criteria:

1. Other malignancy active within the previous 2 years except for basal or squamous cell skin cancer, or CIS of the cervix or breast that has completed curative therapy.
2. Participants with any active autoimmune disease or a documented history of autoimmune disease, except for participants with vitiligo or resolved childhood asthma/atopy
3. Presence of concomitant upper tract urothelial carcinoma or urothelial carcinoma within the prostatic urethra or any other regional/metastatic disease.
4. Known human immunodeficiency virus (HIV) infection.
5. Active infection requiring therapy
6. Major surgery within 4 weeks before the first dose of study drug.
7. Concurrent medical condition requiring the use of immunosuppressive medications or immunosuppressive doses of systemic medications, such as steroids or absorbed topical steroids (doses >10 mg/d prednisone or equivalent).
8. Prolongation of corrected QT (corrected for QTc interval using Frederica's correction factors [QTcF]) interval to >480 millisecond (msec) when electrolytes balance is normal.
9. Significant cardiovascular impairment.
10. Use of illegal recreational drugs.
11. Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin [ß-hCG] (or human chorionic gonadotropin [hCG]) test with a minimum sensitivity of 25 International Units Per Liter (IU/L) or equivalent units of ß-hCG [or hCG]). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
12. Currently enrolled in another clinical study or used any investigational drug or device within 28 days preceding Cycle 1 Day 1 (first dosing day).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2022-09-29 (Estimated); Study Completion 2022-09-29 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation Part: Number of Participants with Dose-limiting Toxicities (DLTs) | Baseline up to 6 weeks of the Induction Cycle (Cycle length is equal to [=] 6 weeks)
  DLTs are any of the toxicities occurring during the 6 weeks of the Induction Cycle and assessed by the investigator as related to study drug. Toxicity will be evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v.5.0).
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline up to 30 days after the last dose of study drug (approximately 42 months)
Dose Expansion Part: Complete Response Rate (CRR) at 3 Months | Up to 3 months
Dose Expansion Part: CRR at 6 Months | Up to 6 months
Dose Expansion Part: CRR at 12 Months | Up to 12 months
Dose Expansion Part: CRR at 18 Months | Up to 18 months
Dose Expansion Part: CRR at 24 Months | Up to 24 months

SECONDARY OUTCOMES:
Dose Escalation Part: CRR at 3, 6, 12, 18 and 24 Months | At Months 3, 6, 12, 18, and 24
DOCR | From the date of first documented CR until the first documentation of confirmed disease recurrence (approximately 42 months)
Local Recurrence Free Rates | At Months 6, 12, 18, and 24
Cmax: Maximum Observed Plasma Concentration for E7766 | Dose Escalation: Induction Phase: Day 1: 0-24 hour post dose; Day 15: 0-8 hour post dose; Maintenance Phase: Cycle 1: Day :0- 8 hours post dose; Dose Expansion: Induction Phase: Day 1, Day 15: 0-8 hour post dose (Cycle length is 3 weeks)
Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for E7766 | Dose Escalation: Induction Phase: Day 1: 0-24 hour post dose; Day 15: 0-8 hour post dose; Maintenance Phase: Cycle 1: Day :0- 8 hours post dose; Dose Expansion: Induction Phase: Day 1, Day 15: 0-8 hour post dose (Cycle length is 3 weeks)
AUC: Area Under the Plasma Concentration Versus Time Curve for E7766 | Dose Escalation: Induction Phase: Day 1: 0-24 hour post dose; Day 15: 0-8 hour post dose; Maintenance Phase: Cycle 1: Day :0- 8 hours post dose; Dose Expansion: Induction Phase: Day 1, Day 15: 0-8 hour post dose (Cycle length is 3 weeks)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - University of Southern California, Los Angeles, California
  - UCLA, Santa Monica, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Indiana University, Indianapolis, Indiana
  - Washington University, St Louis, Missouri
  - The Mount Sinai Hospital, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.